CLINICAL TRIAL: NCT06113510
Title: Non-invasive Coronary Thrombus Imaging to Define the Cause of Acute Myocardial Infarction
Brief Title: Non-invasive Coronary Thrombus Imaging to Define These Cause of Acute Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC23119
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Infarction; Thrombosis
MeSH Terms: conditions — Myocardial Infarction; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples (approximately 20mls)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: 50 patients with myocardial infarction and non-obstructive coronary arteries
  Interventions: Radiation: Hybrid 18F-GP1 positron emission tomography and coronary computed tomography coronary angiography
- 2: 10 patients with suspected coronary thromboembolism 10 patients with suspected spontaneous coronary artery dissection 10 patented with iatrogenic spontaneous coronary artery dissection
  Interventions: Radiation: Hybrid 18F-GP1 positron emission tomography and coronary computed tomography coronary angiography

INTERVENTIONS:
Radiation: Hybrid 18F-GP1 positron emission tomography and coronary computed tomography coronary angiography — 18F-GP1 will be synthesized by our radiochemistry facility, the Edinburgh Imaging Facility Radiochemistry (EIFR), which is co-located within our Edinburgh Imaging Facility, Queens Medical Research Institute (EIF QMRI) using our well-established protocols. Each patient will undergo 18F-GP1 PET/CT coronary angiography imaging on our hybrid scanner (Biograph mCT, Siemens) as soon as practical after their index event and within a maximum of 7 days from symptom onset. Patients will initially be injected with 250 MBq 18F-GP1, before resting in a quiet environment for 60 min. A low-dose attenuation correction CT scan (120 kV, 50 mAs, 5/3 mm) will be followed by acquisition of PET data in list mode using a two 20-min bed position centred on the thoracic aorta and heart. A contrast-enhanced CT coronary angiogram will then be performed.

SUMMARY:
We now have very sensitive blood tests that can pick up damage to the heart and find patients who have had a heart attack. However, whilst this is welcome, it does not identify what causes the heart attack and can sometimes pick up other conditions that cause a strain on the heart.

The classic cause of a heart attack is when a blood clot forms on fatty deposits within the heart arteries. This leads to treating patients with blood thinning medication, and this is very effective and saves lives. However, many apparent heart attacks are not caused by blood clots and some may be caused by blood clots but pass unrecognised.

In this proposal, we will test an exciting new imaging test that can 'see' from outside the body whether there is a blood clot in the heart arteries. This could provide a major new way of assessing patients to ensure they get the right diagnosis and the right treatment. This could ultimately improve the outcomes of or patients with heart attacks.

We will recruit 80 patients in total who have recently been diagnosed with a heart attack from the cardiology department at the Royal Infirmary of Edinburgh. The research team will review patient's medical records to determine eligibility for the study.

The research study involves participants undertaking the following research procedures and assessments:

1. A combined Positron Emission Tomography and Computed Tomography (PET-CT) scan of the heart
2. Ultrasound scan of the heart (Echocardiogram)
3. MRI scan of the heart
4. A blood test - a total of up to four tablespoons (60 mL) of blood will be taken for immediate testing and the remaining blood will be stored for future ethically approved studies
5. A follow up questionnaire 6 -12 months following the heart attack

DETAILED DESCRIPTION:
1.1 BACKGROUND

1.1.1 Background of coronary artery disease and acute myocardial infarction

Coronary artery disease remains the leading cause of death worldwide, with more than 23 million annual deaths estimated to occur by 2030. The introduction of high-sensitivity cardiac troponin measurement has revolutionised the identification and management of patients presenting with acute chest pain and myocardial infarction. However, elevated cardiac troponin concentrations can result from both ischaemic (myocardial infarction) or non-ischaemic (myocardial injury) causes. Moreover, the further subclassification of myocardial infarction relies on the underlying aetiology of infarction which is often not readily apparent and remains a diagnostic challenge.

1.1.2 Universal definition of myocardial infarction

Acute myocardial infarction is defined as cardiomyocyte injury and necrosis in a clinical setting consistent with acute myocardial ischaemia. The fourth universal definition of myocardial infarction describes five subtypes of acute infarction. Type 1 myocardial infarction is characterised by underlying atherosclerotic plaque disruption (rupture, ulceration, fissuring, erosion, or calcific nodules) resulting in intraluminal thrombosis, distal coronary embolisation and intraplaque haemorrhage that ultimately cause myocyte necrosis. In contrast, type 2 myocardial infarction is classified as an ischaemic myocardial injury secondary to oxygen supply and demand mismatch, and importantly is not a consequence of atherosclerotic plaque rupture and coronary atherothrombosis. However, some causes of type 2 myocardial infarction do involve intracoronary thrombus including coronary thromboembolism and spontaneous coronary artery dissection. Currently, invasive coronary angiography remains the primary modality to identify patients presenting with plaque related disruption and coronary thrombosis, ultimately providing the distinction between type 1 and type 2 myocardial infarction. However, it is not always definitive and only 10-20% of patients presenting with type 2 myocardial infarction undergo further investigations to identify the presence of underlying coronary artery disease or to exclude coronary atherothrombosis. Indeed, we recently demonstrated comprehensive cardiac imaging and coronary angiography that identified two thirds of patients had previously unrecognised underlying coronary artery disease, and this resulted in diagnostic reclassification of many patients. These standard techniques were however unable to determine whether this plaque was implicated in the presentation or simply a bystander finding. A non-invasive imaging technique to reliably detect intracoronary thrombus and facilitate this distinction would therefore be of major clinical value.

1.1.3 Imaging intracoronary thrombosis

At present, invasive coronary angiography is the primary modality used to detect the presence of intracoronary thrombus in patients presenting with acute myocardial infarction, through an abrupt occlusion of the coronary artery or a filling defect in partially occluded vessels. This approach has high specificity but low sensitivity for detection of intracoronary thrombus, necessitating the introduction of adjunctive invasive coronary intravascular imaging including angioscopy, intravascular ultrasound and optical coherence tomography to improve rates of identification of coronary thrombosis and atherothrombosis. Intravascular ultrasound-based studies have indicated an incidence of plaque disruption of 30-40% in patients with myocardial infarction and non-obstructive coronary arteries, although this imaging technique cannot differentiate between echo-lucent plaques and acute thrombus. Optical coherence tomography has replaced intravascular ultrasound as the gold standard in high-resolution cross-sectional imaging of the arterial intima, providing a more detailed assessment of coronary artery dissection and thrombus formation. However, these invasive techniques are not always available, have limitations in respect to assessing smaller or stenosed vessels, and only provide circumstantial evidence of the presence of a thrombus based on the characteristic appearances of the images. As such, atherothrombotic events may be missed, resulting in misdiagnosis and, importantly, a missed opportunity to establish patients on appropriate treatment and secondary prevention.

1.1.4 Uncertain role of coronary thrombosis in myocardial infarction

An accurate diagnosis is imperative for establishing subsequent appropriate therapeutic intervention in patients with myocardial infarction. Patients presenting with type 1 myocardial infarction require short-term anticoagulation as well as medium-term dual antiplatelet therapy, in conjunction with other secondary prevention therapies. For most patients with type 2 myocardial infarction, the above strategy would be both ineffective and potentially harmful, such as in patients with bleeding associated anaemia. However, intracoronary thrombus formation underpins certain causes of type 2 myocardial infarction including coronary thromboembolism and spontaneous coronary artery dissection. Accurate identification of intracoronary thrombus is a central tenet in both the diagnosis of type 1 myocardial infarction, and in the differentiation of the various aetiologies underlying type 2 myocardial infarction.

1.1.4.1 Myocardial infarction with non-obstructive coronary arteries

Co-existing coronary artery disease is common in patients with myocardial infarction and non-obstructive coronary arteries, with plaque disruption being the key trigger of acute myocardial infarction in many cases. Myocardial infarction and non-obstructive coronary arteries was first documented over 75 years ago when pathological studies reported evidence of myocardial necrosis in the absence of coronary atherosclerosis. Its recognition in clinical practice remains more recent, and it comprises a heterogenous group of vascular or myocardial disorders, occurring in 5-15% of patients presenting with acute myocardial infarction. Compared to patients with obstructive coronary artery disease, patients with myocardial infarction and non-obstructive coronary arteries are younger, more likely to be female, and have specific genetic and ethnic predispositions. Interestingly, the prevalence of traditional coronary artery risk factors including dyslipidaemia, hypertension and diabetes mellitus is lower in patients with myocardial infarction and non-obstructive coronary arteries.

Myocardial infarction and non-obstructive coronary arteries has defined criteria as outlined by the European Society of Cardiology in 2017 and the American Heart Association/American College of Cardiology in 2019. To fulfil the diagnosis, patients must present with (i) acute myocardial infarction as defined by the fourth universal definition of myocardial infarction, (ii) non-obstructive coronary arteries on angiography (no coronary artery stenosis ≥ 50%), and (iii) no specific alternative diagnosis for the clinical presentation. Only ischaemic causes of acute myocardial infarction are now included in the underlying aetiology of myocardial infarction and non-obstructive coronary arteries. This includes patients presenting with either type 1 or type 2 myocardial infarction but excludes those with takotsubo cardiomyopathy and myocarditis. Although this has simplified the diagnostic work-up of this patient cohort, there remains a high degree of variability in the way patients with suspected myocardial infarction and non-obstructive coronary arteries are investigated and treated, because it is a diagnosis of exclusion. The identification and management of these patients will depend on local practice and resources, where there may be limited access to more advanced diagnostic testing. This is likely one of the contributory factors underlying a recent analysis demonstrating that patients with myocardial infarction and non-obstructive coronary arteries had a higher one-year adjusted mortality than patients with myocardial infarction and obstructive coronary artery disease. As such, there is a clinical need to improve the accuracy in the identification, investigation, and management of this patient population.

1.1.4.2 Coronary thromboembolism

Coronary thromboembolism results in myocardial infarction and non-obstructive coronary arteries if it involves the microcirculation or if the epicardial coronary thrombus is not associated with atherosclerotic coronary artery disease. Underlying aetiologies can range from atrial fibrillation, hypercoagulable states, inherited thrombophilia, paradoxical embolism, valvular vegetations, valvular calcifications and cardiac tumours. As this subtype of event typically involves smaller calibre coronary vessels, their identification using catheter-based techniques is limited by the inability to access smaller vessels due to the size and physical limitations of the intravascular probes. A more sensitive novel and non-invasive imaging modality that can more accurately assess small calibre coronary vessel thrombosis would be of great clinical value to identify coronary thrombosis events resulting in type 2 myocardial infarction.

1.1.4.3 Spontaneous coronary artery dissection

Spontaneous coronary artery dissection is an uncommon cause of acute myocardial infarction, with a predominance in younger (<50 years) women. Myocardial ischaemia is driven by obstruction to coronary blood flow, secondary to separation of medial and adventitial coronary vascular walls, with associated intramural haematoma resulting in protrusion into the coronary arterial lumen. The coronary arteries can appear normal or near normal on coronary angiography, due to gradual tapering of the vessel, and this is commonly a missed diagnosis. Moreover, the prevalence of iatrogenic catheter-induced coronary artery dissection is reported to be increased in patients with spontaneous coronary artery dissection, meaning that many clinicians are reluctant to perform intravascular imaging in patients with this suspected diagnosis. Consequently, the true incidence of spontaneous coronary artery dissection is likely to be underestimated.

1.1.5 Non-invasive imaging of coronary thrombus - Pilot data

We have recently used positron emission tomography (PET) with computed tomography (CT) coronary angiography to identify intracoronary thrombus using a novel radiotracer, 18F-GP1. This radiotracer is highly selective and specific for the activated glycoprotein IIb/IIIa receptor on activated platelets. As part of a previous BHF-funded Clinical Research Training Fellowship (Dr Evangelos Tzolos; FS/CRTF/20/24086) and Project Grant (PG/19/40/34422), we have demonstrated that 18F-GP1 has specificity for the detection of intravascular thrombosis in a range of cardiovascular conditions. We have recently undertaken studies in patients with coronary atherothrombosis in acute type 1 myocardial infarction. This was the first demonstration that non-invasive imaging can identify in vivo intracoronary thrombus in patients presenting with acute myocardial infarction, and for this work, Dr Tzolos was awarded the European Society of Cardiology Young Investigator Award in 2021. We have confirmed the high selectivity and specificity of 18F-GP1 binding to activated platelets within fresh human thrombus and coronary thrombectomy specimens, and importantly we have observed 18F-GP1 uptake only occurs within the culprit coronary arteries of those with acute myocardial infarction. For example, in patients with triple vessel disease, coronary 18F-GP1 uptake was only seen at the site of the culprit lesion. We have also demonstrated preliminary findings of focal 18F-GP1 uptake at the site of spontaneous coronary artery dissection, coronary thromboembolism and extra-coronary thrombus including unrecognized left ventricular and atrial thrombus, as well as infarct-related intramyocardial 18F-GP1 uptake. This changed both the diagnosis (type 1 reclassified as type 2 myocardial infarction) and the treatment (initiation of anticoagulation) of patients presenting with acute myocardial infarction. These data demonstrate the feasibility of identifying patients with intracoronary thrombus and type 1 myocardial infarction, and those with type 2 myocardial infarction caused by spontaneous coronary artery dissection and coronary thromboembolism. Importantly the pattern of 18F-GP1 distribution differs among these three conditions, allowing their differentiation. This technique holds major promise in aiding the classification of myocardial infarction, especially in patients with myocardial infarction and non-obstructive coronary arteries or where the presence of coronary thrombosis is unclear.

1.2 RATIONALE FOR STUDY

With the evolving complexity in modern diagnostic criteria and treatments, it has become increasingly important to determine the aetiology of acute myocardial infarction and specifically determine the presence of intracoronary thrombosis. This has major implications for treatment decisions and patient outcome. However, there are currently no techniques that can reliably determine the presence of intracoronary thrombus throughout the coronary circulation. Here, we will assess a promising highly sensitive and accurate technique to determine the contribution of coronary thrombosis in patients presenting with uncertain or difficult to diagnose causes of myocardial infarction. This will potentially provide a completely novel approach that could provide major insights into the diagnosis, investigation and treatment of these patients.

2 STUDY OBJECTIVES

2.1 OBJECTIVES

2.1.1 Primary Objective The primary objective of this study is to establish the origin, frequency and distribution of activated platelets and thus thrombotic causes of myocardial infarction in patients presenting with myocardial infarction with non-obstructive coronary arteries 2.1.2 Secondary Objectives To inform the pathophysiology and understanding of acute myocardial subtypes, by providing additional mechanistic information regarding the presence of intracoronary activated platelets and thrombosis.

2.2 ENDPOINTS

2.2.1 Primary Endpoint

The primary endpoint will be the degree and location of platelet activation as determined by the target to background ratio of 18F-GP1.

2.2.2 Secondary Endpoints

The secondary endpoints will include measuring the presence of platelet activation in acute myocardial infarction with non-obstructive coronary arteries and identifying the presence and site of platelet activation in thrombosis-related coronary causes of type 2 myocardial infarction.

3 STUDY DESIGN

This will be a prospective observational case-control cohort study

4 STUDY POPULATION

4.1 NUMBER OF PARTICIPANTS

We will recruit two patient populations after invasive coronary angiography has been completed. We have established comparator control populations including 50 patients with stable coronary artery disease (no angina or recent myocardial infarction) and valvular heart disease who underwent 18F-GP1 cardiac PET-CT as part of a concurrent study (NCT04073875) (34).

4.1.1 Cohort 1: Patients with myocardial infarction with non-obstructive coronary arteries

We will recruit 50 patients with myocardial infarction and non-obstructive coronary arteries on coronary angiography

4.1.2 Cohort 2: Patients with coronary causes of type 2 myocardial infarction

We will recruit 10 patients with coronary artery thromboembolism and 10 patients with spontaneous coronary artery dissection. Finally, we will include 10 subjects who have had iatrogenic coronary artery dissection or intramural haematoma as a complication of their percutaneous coronary intervention.

4.2 INCLUSION CRITERIA

* Males and females ≥ 18 years of age
* Clinical presentation of chest pain, ST-segment deviation within a coronary artery territory on the electrocardiogram, raised cardiac troponin and non-obstructive coronary arteries on invasive coronary angiography as per international societal diagnostic criteria (19, 26).

4.3 EXCLUSION CRITERIA

* <18 years of age
* Takatsubo cardiomyopathy
* Myocarditis
* Renal failure (estimated glomerular filtration rate <30 mL/min/1.73 m2)
* Woman of child-bearing potential who are pregnant or breastfeeding
* Known allergy or contraindication to iodinated contrast or radiotracer
* Patients unable to tolerate the supine position
* Patients unable to provide informed consent

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Clinical presentation of chest pain, ST-segment deviation within a coronary artery territory on the electrocardiogram, raised cardiac troponin and non-obstructive coronary arteries on invasive coronary angiography as per international societal diagnostic criteria

Exclusion Criteria:

* <18 years of age
* Takatsubo cardiomyopathy
* Myocarditis
* Renal failure (estimated glomerular filtration rate <30 mL/min/1.73 m2)
* Woman of child-bearing potential who are pregnant or breastfeeding
* Known allergy or contraindication to iodinated contrast or radiotracer
* Patients unable to tolerate the supine position
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit two patient populations after invasive coronary angiography has been completed. We have established comparator control populations including 50 patients with stable coronary artery disease (no angina or recent myocardial infarction) and valvular heart disease who underwent 18F-GP1 cardiac PET-CT as part of a concurrent study (NCT04073875).
  Cohort 1: Patients with myocardial infarction with non-obstructive coronary arteries
  We will recruit 50 patients with myocardial infarction and non-obstructive coronary arteries on coronary angiography
  Cohort 2: Patients with coronary causes of type 2 myocardial infarction
  We will recruit 10 patients with coronary artery thromboembolism and 10 patients with spontaneous coronary artery dissection. Finally, we will include 10 subjects who have had iatrogenic coronary artery dissection or intramural haematoma as a complication of their percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the degree and location of platelet activation as determined by the target to background ratio of 18F-GP1 | 3 years

SECONDARY OUTCOMES:
The secondary endpoints will include measuring the presence of platelet activation in acute myocardial infarction with non-obstructive coronary arteries and identifying the presence and site of platelet activation in thrombosis-related coronary causes of | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Our objective is to non-invasively determine the prevalence of coronary thrombosis in patients presenting with acute myocardial infarction of uncertain aetiology using the novel radiotracer 18F-GP1, and further evaluate its added clinical value in aiding the diagnosis and treatment of these patients.
Supporting Information: Study Protocol, ICF
Time Frame: Resources and timescale: The project will run for 36 months. As principle investigator the majority of this period will involve the recruitment of patients, imaging acquisition and analysis and data analysis. Throughout the project, period publications will be generated with the main publications being generated towards the end of of the study.
Access Criteria: Information will be disseminated internally to the cardiovascular research team through monthly departmental meetings. This will provide an opportunity to update on process, share knowledge with researchers who are also undertaking projects involving 18F-GP1 CT-PET. Communication on a wider scale will be through research publications.

DOCUMENTS (2):
  • Study Protocol (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT06113510/Prot_000.pdf
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT06113510/ICF_001.pdf